CLINICAL TRIAL: NCT06437301
Title: End Tidal CO2 and Masks: Is There a Correlation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Peter Richman, MD, Professor and Research Director, CHRISTUS Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-057
Record Dates: First submitted 2024-03-07; First posted 2024-05-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypercapnia
Keywords: Hypoxia; Respiratory Disease; Surgical Mask; Physiologic Capacity; Oxygen; Sympathetic Nerve Activity
MeSH Terms: conditions — Hypercapnia; Hypoxia; Respiration Disorders | interventions — Masks

STUDY DESIGN:
Intervention Model Description: This study is a prospective, controlled study involving healthy adult volunteers all of whom are resident and faculty physicians, or other medical staff. There will be no financial compensation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline ETCO2 without mask (Other): Subjects will have their baseline end tidal carbon dioxide measured while at rest and without a mask.
  Interventions: Other: Baseline measure of ETCO2 without mask
- Baseline ETCO2 with mask (Other): The second measurement will also occur at rest, but while subjects are wearing a mask.
  Interventions: Other: Baseline ETCO2 with mask
- ETCO2 after 200 meter walk with mask (Other): Lastly, end tidal carbon dioxide will be measured after each participant walks 200 meters, with a surgical mask.
  Interventions: Other: ETCO2 after 200 meter walk with mask
- ETCO2 after 200 meter walk without mask (Other): Lastly, end tidal carbon dioxide will be measured after each participant walks 200 meters, without a surgical mask.
  Interventions: Other: ETCO2 after 200 meter walk without mask

INTERVENTIONS:
Other: Baseline measure of ETCO2 without mask — Baseline
  Arms: Baseline ETCO2 without mask
Other: Baseline ETCO2 with mask — Mask
  Arms: Baseline ETCO2 with mask
Other: ETCO2 after 200 meter walk with mask — 200 meter walk and mask
  Arms: ETCO2 after 200 meter walk with mask
Other: ETCO2 after 200 meter walk without mask — 200 meter walk
  Arms: ETCO2 after 200 meter walk without mask

SUMMARY:
In light of the ongoing COVID-19 pandemic, wearing a mask has become a universal standard as an attempt to reduce the spread of COVID-19. As of 2020, more than half of all U.S. states have implemented a state wide mandated mask policy. There are many schools of thought regarding the benefits and risks of donning a mask to prevent the spread of COVID-19. There is an unproven theory among some that wearing a mask interferes with our natural respiratory function, causing hypoxia, altered mental status and other various health issues. This dangerous perception has led some to believe wearing a mask is harmful, and encourages against wearing a mask in public. This theory, recently refuted by a study investigating oxygen levels while participants wore masks, performed in 2020 encouraged increased compliance with wearing masks. Another study, preformed by evaluated whether gas exchange abnormalities occurred with the use of surgical masks in subjects with and without lung function impairment. The conclusions of the study showed that regardless of lung function impairment, the presence of surgical masks did not impact gas exchange. Additionally, a more recent study concluded that the presence of a facemask did not have a significant change in physiologic parameters while during exercise. Although there is evidentiary support that facemasks do not negatively affect oxygen status and physiologic capacity, there is not strong evidence examining the relationship between ETCO2 and facemasks. The relationship between ETCO2 and facemasks is one of importance because mild decreases in oxygen have much less dangerous effects compared to the effects of rapid accumulations of carbon dioxide. Increases in end tidal carbon dioxide lead to confusion, acidosis and in severe cases, respiratory distress and failure. A study performed in 1989 showed that hypercapnia has greater increases in blood pressure, minute ventilation and sympathetic nerve activity than hypoxia.

In this newly proposed study, healthy volunteers will all wear the same type of three layer surgical mask. Their end tidal carbon dioxide will be measured while at rest without a mask, while resting with a mask and then after walking 100 meters in the mask. While previous studies have focused on changes in oxygen, there is a lack of research dedicated to analyzing end tidal carbon dioxide. This study will hope to show evidence supporting that there is no increase in end tidal carbon dioxide while wearing a mask.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18 and 75
* Consent to participate in this study
* Resident and ancillary staff

Exclusion Criteria:

* Patients
* Inability or refusal consent
* Inability to walk the predetermined distance
* History of lung disease
* History of significant cardiac disease
* People under the age of 18 and over the age of 75

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Change in end tidal carbon dioxide while wearing a mask. | Measured immediately after mask was put on.
  The primary objective of this study is to evaluate if there are changes present with non-invasive end tidal carbon dioxide measurement while wearing a mask.

SECONDARY OUTCOMES:
Change in end tidal carbon dioxide while wearing a mask and walking a moderate distance. | Measured a time = 0 seconds after walk was completed.
  The secondary objective is to assess possible changes in end tidal carbon dioxide while walking moderate distances (200 meters) while wearing a mask.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRISTUS Health-Texas A&M Spohn Emergency Medicine Residency, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan NC, Li K, Hirsh J. Peripheral Oxygen Saturation in Older Persons Wearing Nonmedical Face Masks in Community Settings. JAMA. 2020 Dec 8;324(22):2323-2324. doi: 10.1001/jama.2020.21905. PMID 33125030
- [Result] Barbeito-Caamano C, Bouzas-Mosquera A, Peteiro J, Lopez-Vazquez D, Quintas-Guzman M, Varela-Cancelo A, Martinez-Ruiz D, Yanez-Wonenburger JC, Pineiro-Portela M, Vazquez-Rodriguez JM. Exercise testing in COVID-19 era: Clinical profile, results and feasibility wearing a facemask. Eur J Clin Invest. 2021 Apr;51(4):e13509. doi: 10.1111/eci.13509. Epub 2021 Feb 15. PMID 33548060
- [Result] Samannan R, Holt G, Calderon-Candelario R, Mirsaeidi M, Campos M. Effect of Face Masks on Gas Exchange in Healthy Persons and Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2021 Mar;18(3):541-544. doi: 10.1513/AnnalsATS.202007-812RL. No abstract available. PMID 33003954
- [Result] Somers VK, Mark AL, Zavala DC, Abboud FM. Contrasting effects of hypoxia and hypercapnia on ventilation and sympathetic activity in humans. J Appl Physiol (1985). 1989 Nov;67(5):2101-6. doi: 10.1152/jappl.1989.67.5.2101. PMID 2513316
- See also: What U.S. States Require Masks In Public? — https://masks4all.co/what-states-require-masks/
- See also: Adverse Effects of Prolonged Mask Use among Healthcare Professionals during COVID-19 — http://clinmedjournals.org/articles/jide/journal-of-infectious-diseases-and-epidemiology-jide-6-130.php?jid=jide

DOCUMENTS (1):
  • Study Protocol (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT06437301/Prot_000.pdf